CLINICAL TRIAL: NCT01357317
Title: Changes in Biochemical and Vascular Parameters w/Lanthanum Carbonate & Calcium Acetate Therapy Compared to Dietary Intervention in Pts w/Stage 3 & 4 Chronic Kidney Disease & Abnormal Phosphorus Homeostasis: a Randomized Controlled Trial
Brief Title: Study Comparing Effects of Lanthanum Carbonate Versus Calcium Acetate Versus Dietary Phosphorus Restriction
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Salem Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: Shire (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CK 0036
Record Dates: First submitted 2011-04-04; First posted 2011-05-20 (Estimated); Last update posted 2012-06-12 (Estimated); Status verified 2011-04

CONDITIONS: Chronic Kidney Disease
Keywords: Kidney disease; Hyperphosphatemia; Parathyroid hormone
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Diseases; Hyperphosphatemia | interventions — calcium acetate; lanthanum carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Lanthanum Carbonate (Active Comparator): Lanthanum Carbonate: initial dose 500 mg TID with meals, titrated at monthly intervals in 500 mg increments or decrements, with goal of returning to normal the level of the abnormal baseline marker(s) of phosphorus homeostasis (serum phosphorus, PTH or TRP). Normality for this marker will be defined as serum phosphorus of 2.6-4.6 mg/dl, PTH of 10-65pg/ml and TRP>=80%.
  Interventions: Other: Diet counseling
- Calcium Acetate (Active Comparator): Calcium Acetate: initial dose 667 mg TID with meals, titrated at monthly intervals in 667 mg increments or decrements, with goal of returning to normal the level of the abnormal baseline marker(s) of phosphorus homeostasis. The maximum daily intake of elemental calcium should not exceed 1500 mg in order to comply w/recommendations from K-DOQI [5](this is approximately equal to three 667mg tablets of calcium acetate TID).
  Interventions: Other: Diet counseling
- Dietary instructions (Active Comparator): Dietary instructions consisting of pamphlets describing foods high in phosphorus and consultation with a renal dietitian if necessary, with the goal of return to normal the level of the abnormal marker of phosphorus homeostasis. Rescue therapy with a phosphorus binder of the treating physician's choice will be allowed in patients who fail to normalize elevated baseline serum phosphorus levels after 3 months following dietary instructions.
  Interventions: Drug: Phosphorus binder

INTERVENTIONS:
Other: Diet counseling — If serum phosphorus level exceeds 4.6 mg/dl in the lanthanum carbonate arm in spite of consecutive up-titration of the medical dose or due to patients' intolerance of the medication, patient will be considered a treatment failure and other treatment options will be implemented, including diet counseling or another class of phosphorus binder (in this order of preference).
  Other Names: calcium acetate
  Arms: Lanthanum Carbonate
Other: Diet counseling — If serum phosphorus level exceeds 4.6 mg/dl in spite of consecutive up-titration of the medication dose or due to patients' intolerance of the medication, patient will be considered a treatment failure and other treatment options will be implemented, including diet counseling or another class of phosphorus binder (in this order of preference).
  Other Names: Lanthanum Carbonate
  Arms: Calcium Acetate
Drug: Phosphorus binder — If serum phosphorus level exceeds 4.6 mg/dl after 3 months of concerted efforts, the patient will be considered a treatment failure and treatment with a phosphorus binder of the treating physician's choice will be allowed.
  Other Names: Lanthanum Carbonate; Calcium Acetate
  Arms: Dietary instructions

SUMMARY:
Objective: To examine the effects of three commonly applied treatments of disordered phosphorus homeostasis on biochemical markers and vascular characteristics in patients with moderate and advanced non-dialysis dependent chronic kidney disease.

DETAILED DESCRIPTION:
Approximately 120 qualified patients from our medical center, who have been diagnosed with mild to moderate chronic kidney disease (estimated GFR 15-60 ml/min), will be enrolled. After informed consent, qualified subjects will be randomized into 3 arms in a 1:1:1 ratio: lanthanum carbonate, calcium acetate, and dietary modification. The maximum length of treatment is 12 months. Dose of intervention will be adjusted based on changes in biochemical parameters. Primary end points are changes in serum phosphorus, urine phosphorus, serum parathyroid hormone, coronary artery calcification, aortic pulse velocity and flow mediated vasodilation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female CKD patients > 18 years old
* Patients should be willing and able to provide written informed consent and HIPAA authorization to participate in study
* Chronic kidney disease Stage 3 or 4 per K-DOQI Guidelines: estimated glomerular filtration rate (eGFR) of 15-60 ml/.min/1.73m2 by using modified MDRD equation.
* Serum phosphorus >4.6 mg/dl or plasma intact PTH (iPTH) level above 65 pg/ml or tubular reabsorption of phosphorus (TRP) <80%.
* A negative pregnancy test prior to enrollment in female patients, unless the patient is 2 years postmenopausal, or has had a documented tubal ligation or total hysterectomy.
* Patients need to be off any phosphorus binders for 4 weeks prior to screening
* Stable dose of vitamin D products for 4 weeks in patients receiving such agents. Dose changes in patients receiving stable and initiation of vitamin D products in patients previously not treated will not be permitted during study

Exclusion Criteria:

* Women who are pregnant, capable of becoming pregnant and not participating in an acceptable form of birth control, or who are breast feeding
* Patients currently participating in a clinical trial with another investigational drug or device or who have receiving an investigational drug or device within 30 days of enrollment in this study
* Major surgery within 2 month prior to enrollment in study or planned surgery while the patient is in the study, other than dialysis vascular access surgery.
* Presence of coronary stents, artificial heart valves or pacemakers, and history of CABG
* Patients with active infections requiring ongoing treatment
* Patients who have had a malignancy (except for non-melanoma cancer of the skin) unless the patient has received curative treatment and has been disease free for >2 years
* Patient who the Investigator determines has a medical status that would preclude the patient's participation in the study
* Patients on hemodialysis (HD) or peritoneal dialysis (PD)
* Patients with a functional renal transplant
* Patients with allergies to study drugs
* Patients with serum calcium >10.7 mg/dl.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2011-06; Primary Completion 2013-10 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Designated safety measure; serum calcium | 1 year compared to day 0
  Changes in calcium, PTH, FGF-23 at 1 year compared to day 0
Designated safety measure: phosphorus | 1 year compared to day 0
  Changes in serun phosphorus, tubular reabsorption of phosphorus, bone-specific alkaline phosphatase at 1 year compared to day 0

SECONDARY OUTCOMES:
Changes in flow | 1 year compared to day 0
  Changes in flow mediated vasodilatation at 1 year compared to day 0.
Other Changes | 1 year compared to day 0
  Changes in pulse wave velocity, central aortic blood pressure, coronary artery calcification at 1 year compared to day 0.

CONTACTS AND LOCATIONS:
Overall Officials: Csaba P. Kovesdy, M.D., Principal Investigator — Salem VAMC
Locations (1):
- VA Medical Center, Salem, Virginia, United States

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086
- [Derived] Kovesdy CP, Lu JL, Wall BM, Gyamlani G, Naseer A, Wallick A, Han Z, Thomas F, Quarles LD, Jarmukli N. Changes With Lanthanum Carbonate, Calcium Acetate, and Phosphorus Restriction in CKD: A Randomized Controlled Trial. Kidney Int Rep. 2018 Mar 23;3(4):897-904. doi: 10.1016/j.ekir.2018.03.011. eCollection 2018 Jul. PMID 29989014